CLINICAL TRIAL: NCT06804460
Title: Effect of a Vegan Mediterranean Diet on Cardiometabolic Biomarkers, Functional Capacity, and Quality of Life in Patients with Fibromyalgia
Acronym: FIBROVEG
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Miguel López Moreno, Principal Investigator, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGL-2024-46 project
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vegan Mediterranean diet (Experimental): The vegan mediterranean diet is mainly composed of whole plant-based foods, similar to a Mediterranean diet, but the animal sources of protein and fat are substituted with plant foods rich in protein and fat. During the vegan diet, participants are supplemented with 1000 µg of cyanocobalamin (vitamin B12) twice a week (Harrison Sports Nutrition, Granada, Spain) to compensate for the deficiency in vitamin B12 intake induced by the vegan diet.
  Interventions: Behavioral: Dietary intervention
- Mediterranean diet (Active Comparator): The traditional Mediterranean diet contains an abundant intake of whole plant-based foods, with moderate to low consumption of fish, poultry, low-fat dairy products, and eggs, very low consumption of red and processed meats, and no sweets. Olive oil is the main added fat, and animal protein accounts for 60% of total protein intake.
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — The vegan mediterranean diet is mainly composed of whole plant-based foods, similar a una dieta mediterránea, but the animal sources of protein and fat are substituted with plant foods rich in protein and fat. During the vegan diet, participants are supplemented with 1000 µg of cyanocobalamin (vitamin B12) twice a week (Harrison Sports Nutrition, Granada, Spain) to compensate for the deficiency in vitamin B12 intake induced by the vegan diet.

SUMMARY:
This study aims to evaluate the effect of a vegan Mediterranean diet compared to a traditional Mediterranean diet on inflammatory biomarkers, functional capacity, and quality of life in patients with fibromyalgia.

DETAILED DESCRIPTION:
The study involves two visits to the Exercise Physiology Research Laboratory at UFV. During the first visit, participants will complete functional capacity tests, respond to questionnaires (Fibromyalgia Impact Questionnaire, Short Form-36, MDF-Fibro-17, and Tampa Scale for Kinesiophobia), and provide a blood sample from the antecubital vein collected by an auxiliary nurse from the Eurofins MEGALABS laboratory. The biochemical markers to be analyzed include: white blood cell count (neutrophils, lymphocytes, monocytes, and platelets), lipid profile, fasting blood glucose levels and acute-phase proteins (C-reactive protein). Additionally, body composition will be assessed using a Tanita TBF300, and waist circumference will be measured. Functional capacity tests will include a handgrip strength test, a 30-second chair-to-stand test, and a timed up-and-go test. Participants will undergo a six-week dietary intervention and will return for a second visit at the end of the intervention period. They will be randomly assigned to follow either a vegan Mediterranean diet or a traditional Mediterranean diet, both of which will be guided and supervised by registered dietitians. These diets will be designed to meet individual energy needs and key nutrient requirements, following the standards set by the National Academy of Medicine and the Academy of Nutrition and Dietetics. Both diets will be isocaloric and maintain an identical macronutrient distribution. After the intervention, participants will repeat the same functional tests, questionnaires, and capillary blood measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 50 years.
* Participants with a Fibromyalgia diagnosis according to the American College of Rheumatology (ACR) criteria.
* Functional independence.
* Non-smokers.
* Low alcohol consumption (<1 serving/day).
* Pharmacological treatment stabilized for at least 4 weeks prior to the start of the study.

Exclusion Criteria:

* Pregnant, lactating, or menopausal women.
* Physical condition that prevents the performance of functional capacity tests.
* Change in pharmacological therapy during the intervention period.
* Concomitant inflammatory conditions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-04-14 (Estimated); Study Completion 2025-04-21 (Estimated)

PRIMARY OUTCOMES:
Neutrophil to lymphocyte ratio | From enrollment to the end of treatment at 6 weeks
  Lymphocyte and neutrophil concentrations will be measured with the HemoCue® WBC DIFF system (HemoCue AB, Ängelholm, Sweden).The Neutrophil-to-Lymphocyte Ratio (NLR) is a simple inflammatory biomarker calculated by dividing neutrophil count by lymphocyte count. It reflects the balance between inflammation (neutrophils) and immune regulation (lymphocytes).
  An elevated NLR is associated with chronic inflammation, physiological stress, or immune dysfunction, while lower levels indicate a more balanced immune state. Its ease of measurement and broad applicability make it valuable for monitoring inflammatory, cardiovascular, and oncological conditions.
Lipid profile | From enrollment to the end of treatment at 6 weeks
  The concentrations of total cholesterol and cholesterol-LDL will be measured with a POC multi-parameter lux meter (Biochemical Systems International, Italy).
Cardiorespiratory fitness | From enrollment to the end of treatment at 6 weeks
  The 30s Chair-to-Stand (CS) test assesses lower trunk strength by counting how many times a person can stand up and sit down within 30 seconds. It is commonly used to evaluate functional mobility and endurance in older adults or individuals with certain health conditions.
Quality life | From enrollment to the end of treatment at 6 weeks
  The Fibromyalgia Impact Questionnaire (FIQ) examines the impact of fibromyalgia on daily life, covering areas such as functional capacity, pain, fatigue, sleep, and psychological well-being. Its revised version (FIQ-revised) focuses more on functional capacity, symptoms, and the overall impact of fibromyalgia on the individual's daily life.
Metabolic health | From enrollment to the end of treatment at 6 weeks
  Visceral fat is the fat stored within the abdominal cavity around internal organs. It is commonly measured to assess the risk of metabolic diseases, such as type 2 diabetes and cardiovascular conditions.

SECONDARY OUTCOMES:
Metabolic health | From enrollment to the end of treatment at 6 weeks
  Fasting blood glucose measures the level of glucose in the blood after an overnight fast. It is used to assess insulin sensitivity and diagnose conditions like diabetes or prediabetes.
Metabolic health | From enrollment to the end of treatment at 6 weeks
  Triglycerides are a type of fat (lipid) found in the blood, and their concentration is measured to assess cardiovascular health. High levels of triglycerides can increase the risk of heart disease and other metabolic conditions.
Strength performance | From enrollment to the end of treatment at 6 weeks
  handgrip strength test evaluate the strength of the hand and forearm muscles. It is commonly used as an indicator of overall muscle strength and functional capacity.
Quality Life | From enrollment to the end of treatment at 6 weeks
  The Tampa Scale for Kinesiophobia (TSK) will assess the degree of fear of movement or re-injury in individuals with pain or injury. The scale ranges from 17 (minimum) to 68 (maximum) points, with higher scores indicating a worse outcome, as they reflect greater fear of movement or re-injury. This tool helps understand how fear of movement can affect recovery and physical function.
Quality life | From enrollment to the end of treatment at 6 weeks
  The Pittsburgh Sleep Quality Index assesses the quality and patterns of sleep over a one-month period. It is commonly used to evaluate sleep disturbances and their impact on overall health and well-being.

IPD SHARING:
Plan to Share IPD: No
In our study, the sharing of individual participant data (IPD) is not required as part of the trial registration process on ClinicalTrials.gov. The study does not involve sharing identifiable participant information or IPD for secondary analyses or public access